CLINICAL TRIAL: NCT02776293
Title: Prenatal Listening to Songs Composed for Pregnancy and Symptoms of Anxiety and Depression: a Pilot Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Goldsmiths, University of London (Other)
Responsible Party: Principal Investigator, Lauren Stewart, Dr. Lauren Stewart, Goldsmiths, University of London
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LV-001
Record Dates: First submitted 2016-05-12; First posted 2016-05-18 (Estimated); Last update posted 2017-05-04 (Actual); Status verified 2017-05

CONDITIONS: Prenatal Anxiety; Depression
MeSH Terms: conditions — Depression | interventions — Music Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Relaxation Group (Active Comparator): The relaxation group was asked to listen to their assigned audio file for at least 20 minutes a day and to record each time they had engaged in this activity. The audio file consisted of a two minute introduction. Following this, participants were instructed to sit undisturbed for 20 minutes.
  Interventions: Behavioral: Relaxation
- Music Group (Experimental): The music group was asked to listen to their assigned audio file for at least 20 minutes a day and to record each time they had engaged in this activity. The audio file consisted of a two minute introduction. Following this, participants were instructed to listen to pre-recorded songs specifically composed for pregnancy.
  Interventions: Behavioral: Music

INTERVENTIONS:
Behavioral: Relaxation
  Arms: Relaxation Group
Behavioral: Music
  Arms: Music Group

SUMMARY:
Prenatal anxiety and depression are distressing for the expectant mother and can have adverse effects on her fetus and child. This study aimed to determine whether listening to specially composed songs would be an effective intervention for reducing symptoms of prenatal anxiety and depression over a period of 12 weeks.

DETAILED DESCRIPTION:
Prenatal anxiety and depression has negative implications for both the mother and the developing child, including developmental disorders, low birth weight, and altered immune function. It is therefore very important both to detect and to help ameliorate symptoms of anxiety and depression in pregnant women. Many women do not want pharmacological interventions at this time, and with less severe symptoms it may not be appropriate. Thus there is a need to find non-pharmacological methods of intervention. Psychological therapies such as cognitive behavioural therapy or interpersonal therapy can be effective. But these are often not available for the large numbers of women who could benefit. Though there has been evidence that music has the ability reduce anxiety, no study has quantitatively measured prenatal anxiety and depression over a long period of time. Proof of efficacy could justify investment into music as an inexpensive, and non-stigmatizing method to reduce prenatal anxiety and depression and therefore benefit both the mother and child.

ELIGIBILITY:
Inclusion Criteria:

* English speaking women
* At least 18 years of age.

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 223 (Actual)
Dates: Start 2014-01; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
State-Trait Anxiety Inventory | 12 weeks
  Questionnaire measuring an individual's general level of anxiety (trait) and an individual's anxiety level at the time of taking the questionnaire (state).
Edinburgh Postnatal Depression Scale | 12 weeks
  Questionnaire measuring symptoms of maternal depression

CONTACTS AND LOCATIONS:
Overall Officials: Lauren Stewart, MSc. PhD., Principal Investigator — Goldsmiths, University of London; Centre for Music in the Brain, Department of Clinical Medicine, Aarhus University & The Royal Academy of Music

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Nwebube C, Glover V, Stewart L. Prenatal listening to songs composed for pregnancy and symptoms of anxiety and depression: a pilot study. BMC Complement Altern Med. 2017 May 8;17(1):256. doi: 10.1186/s12906-017-1759-3. PMID 28482901